CLINICAL TRIAL: NCT06481761
Title: The Effectiveness of Double-slot Brackets Versus Single-slot Brackets on the Rate of Canine Retraction: A Randomized Clinical Trial
Brief Title: The Effectiveness of Double-slot Brackets Versus Single-slot Brackets on the Rate of Canine Retraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Raghad Mohsen Ghoneim, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Orth3-3-2
Record Dates: First submitted 2024-06-24; First posted 2024-07-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Rate of Canine Retraction
Keywords: canine retraction; double slot brackets; Orthodontic tooth movement

STUDY DESIGN:
Intervention Model Description: study is a randomized clinical trial, single-center, parallel group, two-arms with 1:1 allocation ratio
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, neither participants nor investigators can be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-slot brackets (Active Comparator): Bonding of the upper arch up to second molars with Roth prescription 0.022x.028" single slot brackets (MINI MS-American orthodontics)
  Interventions: Device: Single-slot brackets
- Double-slot brackets (Experimental): Double slot brackets (SORTECH-South Orthodontic Technology) will be Bonded on the upper arch up to the second molars. The brackets are of Roth prescription & have two slots, cervical 0.018x.025" slot and incisal/occlusal 0.022x.028" slot
  Interventions: Device: Double-slot brackets

INTERVENTIONS:
Device: Double-slot brackets — Miniscrews will be inserted in the buccal alveolar bone between first and second molars bilaterally and ligated to second premolar.
  Canine Retraction using Nickel titanium closed-coil springs delivering a force of 150 gram, extending the spring between the canine and first molar hooks.
  retraction on double 0.016'' Stainless steel round wires in both slots of the double slot brackets.
  Re-activation of the coil spring will be done in the follow up visits to maintain a constant force through the study.
  Arms: Double-slot brackets
Device: Single-slot brackets — Miniscrews will be inserted in the buccal alveolar bone between first and second molars bilaterally and ligated to second premolar.
  Canine Retraction using Nickel titanium closed-coil springs delivering a force of 150 gram, extending the spring between the canine and first molar hooks.
  retraction on single 0.017x0.022'' Stainless steel wire. Re-activation of the coil spring will be done in the follow up visits to maintain a constant force through the study.
  Arms: Single-slot brackets

SUMMARY:
The aim of this Randomized clinical trial is to compare the efficacy of the double slot brackets compared to single slot-brackets in producing a controlled rate of upper canine retraction into premolar extraction space.

patients will be randomly divided into one of the two groups, CBCT (cone beam computed tomography) and dental models will be taken for each patient Pre-retraction and following the study completion.

The rate of retraction will be evaluated for both groups as well as Amount of canine root movement and molar anchorage loss will be also assessed.

DETAILED DESCRIPTION:
Eligible patients will be examined for fulfilling the inclusion criteria. All the recruited patients need extraction of upper first premolars followed by canine retraction with maximum anchorage.

The patients will be randomly allocated to one of the two groups; either Double slot brackets or single slot-brackets group.

In Double slot bracket group, Canine retraction will be made on two 0.016'' StSt (stainless steel) round wires, each in one of the slots of the double slot brackets. while in single slot-bracket group, Retraction will be made on one 0.017''×0.025'' rectangular StSt arch wire .

The patients will be seen on a monthly basis for follow up visit for reactivation of retraction to maintain constant force during the study. An impression will be taken for the patients every visit, fabricated dental models will be digitally scanned. The scanned models will be used to monitor the rate of canine retraction.

Every patient will be asked to take a CBCT image of the upper arch pre Retraction and after the completion of study duration (3 months). After data collection, assessors will carry on the measurements blindly. Statistical analysis of the data will be done and the results will be compared to evaluate the effectiveness of both techniques for canine retraction.

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene.
* Adult Male or Female patients with an age range of 16-26 years old.
* Full set of permanent dentition(excluding third molar).
* Any kind of malocclusion requiring first premolar extraction and canine retraction.
* Patients with type/pattern of crowding that allows leveling and alignment before premolar extraction

Exclusion Criteria:

* History of previous orthodontic treatment.
* Craniofacial deformity.
* Systematic disease or administrating drugs affecting tooth movement.
* Poor oral health.

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
rate of canine retraction | 3 months
  millimeters through superimposed digital models taken for each patient monthly at the follow up visits.

SECONDARY OUTCOMES:
Amount of canine root movement | 3 months
  millimeters through pre and post retraction CBCT (cone beam computed tomography) images of the upper arch
Molar cusp anchorage loss | 3 months
  millimeters through superimposed digital models taken for each patient monthly at the follow up visits. and pre and post retraction CBCT images

CONTACTS AND LOCATIONS:
Overall Officials: Amr R El Beialy, Assoc.Prof, Study Chair — Orthodontic department, Faculty of Dentistry, Cairo University; Nada O El Zawahry, lecturer, Study Director — Orthodontic department, Faculty of Dentistry, Cairo University; Noha A El Ashmawi, lecturer, Study Director — Orthodontic department, Faculty of Dentistry, Cairo University
Locations (1):
- Cairo University, Giza, Egypt